CLINICAL TRIAL: NCT03378804
Title: Randomized Comparison of Two Application Procedures: Programmed Intermittent Epidural Bolus in Patient-controlled Epidural Analgesia (PCEA) Versus Continous PCEA in Abdominal Oncological Surgery
Brief Title: PIEB-PCEA vs CEI-PCEA for Abdominal Oncological Surgery. A Randomized Prospective Clinical Trial
Acronym: PIEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Lara Maria Prien, Research Associate, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: nklnk
Record Dates: First submitted 2017-10-06; First posted 2017-12-20 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Pain, Postoperative
Keywords: PCEA; PIEB; epidural analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PIEB-PCEA (Experimental): Programmed intermittent epidural bolus (PIEB) application of ropivacaine 0.2% with patient-controlled epidural analgesia:
  The background rate is set at 6ml per hour. The patient-controlled bolus function is programmed with 4ml at a lock-out interval of 30min.
  Interventions: Procedure: Programmed intermittent epidural bolus application (PIEB)
- CEI-PCEA (Active Comparator): Continous epidural analgesia with patient-controlled analgesia using ropivacaine 0.2%:
  The background rate is set at 6 ml / h continuously. The patient-controlled bolus function is programmed in with 4ml at a lock-out interval of 30min.
  Interventions: Procedure: Continous epidural analgesia

INTERVENTIONS:
Procedure: Programmed intermittent epidural bolus application (PIEB) — Instead of a continuous background infusion of 6ml/h, one bolus injection is performed at the same amount per hour.
  Arms: PIEB-PCEA
Procedure: Continous epidural analgesia
  Arms: CEI-PCEA

SUMMARY:
The aim of the study is to compare programmed intermittent bolus application and continuous epidural infusion with regard to additionally applied patient-controlled volume of local anesthesia and quality of analgesia.

DETAILED DESCRIPTION:
Usually, patient controlled epidural analgesia (PCEA) is performed with a constant background infusion and patient-controlled bolus applications. An alternative approach is to give boluses at a regular rate for basic medication, instead of the continuous background infusion, maintaining the same amount of medication delivered per hour, (Programmed Intermittent Epidural Bolus injection; PIEB). In both cases, the patient has the option to trigger additional boluses. PIEB has been applied successfully in pain relief for lumbar epidural anesthesia in obstetrics, with better quality of analgesia and less total volume of local anesthetic required. It is assumed that the higher pressure in the epidural space with bolus injection results in a better and more uniform spread of the local anesthetic. In this study the PIEB-mode will be applied in major gynecological and abdominal surgery. In order to address the possibility that the different types of surgery result in different degrees of postoperative pain, the patients are stratified in three groups and randomized within these groups (Wertheim, Whipple, major colon surgery).

ELIGIBILITY:
Inclusion Criteria:

* Abdominal tumors in gynecology and general surgery
* Enlightenment and written consent to the investigation

Exclusion Criteria:

* refusal to participate
* pregnancy and breast feeding period
* general contraindications for thoracic epidural anesthesia (e.g. coagulation disorders, --anticoagulation according to the guidelines of DGAI)
* Impossibility to place the epidural catheter correctly
* Known allergy to the drugs used in the study
* Lack of understanding how to use the patient-controlled system
* postoperative follow-up respiratory assistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-01; Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
Number of additional patient-controlled bolus of ropivacaine 0.2% (consumption in ml) | Beginning of operation -6 pm on the second postoperative day
  The patient-controlled bolus function is programmed with 4ml at a lock-out interval of 30min. The number of additional patient-controlled boli will be read off the epidural pump at 6 pm on the day of surgery, 6 pm on the 1st day and 6 pm on the 2nd day

SECONDARY OUTCOMES:
quality of analgesia | At 6 pm on the day of surgery, 6 pm on the 1st day and 6 pm on the 2nd day
  Measured on a visual analog scale of 0-10 (0="no pain" ; 10= "worst imaginable pain"

OTHER OUTCOMES:
Necessity of additional rescue medication | Beginning of operation until 6 pm on the second postoperative day
  Piritramid 7,5mg
Sensory blockade | Beginning of operation -6 pm on the second postoperative day
  Sensory blockade is measured with a tiptherm, motor blockade on the Bromage scale 0-3 (0= no blockade; 1=Inability to lift legs stretched; 2=Inability to bend knees, 3=Inability to move feet )
Patient satisfaction with pain management | At 6 pm on the day of surgery, 6 pm on the 1st day and 6 pm on the 2nd day
  Measured on a visual analog scale of 0-10
first defecation/flatus | after the operation till the end of hospital stay (max 20days)
  dichotomous yes/no
motor blockade | Beginning of operation -6 pm on the second postoperative day
  motor blockade is measured on the Bromage scale 0-3.

CONTACTS AND LOCATIONS:
Locations (1):
- Philipps Universität Marburg, Marburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wiesmann T, Hoff L, Prien L, Torossian A, Eberhart L, Wulf H, Feldmann C. Programmed intermittent epidural bolus versus continuous epidural infusion for postoperative analgesia after major abdominal and gynecological cancer surgery: a randomized, triple-blinded clinical trial. BMC Anesthesiol. 2018 Oct 30;18(1):154. doi: 10.1186/s12871-018-0613-6. PMID 30376810